CLINICAL TRIAL: NCT02256319
Title: Effects of Dexmedetomidine vs Propofol on the Recordings of Deep Brain Activity (Local Field Potentials) Measured Through Implanted Stimulators
Brief Title: Dexmedetomidine vs Propofol on the Recordings of Deep Brain Activity Measured Through Implanted Stimulators
Acronym: DEXPROPAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DEXPROPAR
Record Dates: First submitted 2014-09-30; First posted 2014-10-03 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-02

CONDITIONS: Parkinson's Disease
Keywords: Deep brain stimulation; Dexmedetomidine; Propofol
MeSH Terms: conditions — Parkinson Disease | interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dexmedetomidine recording (Experimental): Recording registered through the deep brain stimulation electrodes with dexmedetomidine at 0.2 μg/kg/h.
  Interventions: Drug: Dexmedetomidine
- Propofol recording (Active Comparator): Recording registered through the deep brain stimulation electrodes with propofol at plasmatic levels of 0.5, 1, 1.5, 2, 2.5 μg/mL.
  Interventions: Drug: Propofol
- Basal recording (No Intervention): Recording registered through the deep brain stimulation electrodes with no sedation .

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive a loading dose of 1 µg/kg in 10 min before starting the surgery. The maintenance dose will be 0.2-1 µg/kg/h for a Ramsey Sedation Score of 3-4 during the surgery´s preparation. It will be reduced to 0.2 µg/kg/h 15 min before starting the microelectrode recording for a Ramsey Sedation Score of 2. After the placement of the deep brain stimulator we will record the local field potentials activity. In addition, the subscales of rigidity, tremor and bradykinesia of the Unified Parkinson's Disease Rating Scale (UPDRS-III) score will be evaluated. Once the deep brain stimulator recording and neurologic exploration will be over patients will receive a maintenance dose 0.2-1 µg/kg/h until the end of the surgery. It will be stopped to transfer the patient to the ICU.
  Other Names: (S)-4-[1-(2,3-Dimethylphenyl)ethyl]-3H-imidazole
  Arms: Dexmedetomidine recording
Drug: Propofol — The target doses are 0.5, 1, 1.5, 2 and 2.5 µg/kg. For its administration we will use the TCI (target controlled infusion) system. After programming each dose we will wait until the plasma and brain concentration of propofol are stabilized in this target and then we will record the local field potentials activity through the DBS. In addition, the subscales of rigidity, tremor and bradykinesia of the UPDRS-III score will be evaluated.
  Other Names: 2,6-diisopropylphenol
  Arms: Propofol recording

SUMMARY:
This clinical trial has been designed to study and compare changes in deep brain activity (field potentials) in Parkinson's disease (PD) patients while awake, and during sedation with dexmedetomidine or propofol. The recording is made through a deep brain stimulation (DBS) electrode implanted for PD management.

The investigators hypothesize that dexmedetomidine produces fewer changes as compared to propofol, and that those changes are consistent and recognizable when compared to activity in patients not exposed to any sedation. Typification of those changes would in the future allow for patients to undergo this surgery comfortably while not compromising the quality of the recording and of the final clinical outcome. The principal variable analyzed is the signal's power in each of the frequency bands, absolute and relative. The analysis will include usual clinical methods such as rapid Fourier transform (FFT) and window fast Fourier transform (WFFT), wavelet analysis, Gabor, and coherence.

DETAILED DESCRIPTION:
Comparative clinical trial, non blinded, controlled and sequential, evaluating the effects of propofol and dexmedetomidine in the basal ganglia of PD patients through a DBS electrode.

It is a phase IV clinical trial evaluating the effects of a drug outside the approved.

The study takes part in three phases:

1. DBS placement under sedation with dexmedetomidine at 0.2 μg/kg/h. This will be called "dexmedetomidine record".
2. Four days later and with no sedation, a recording will be registered in one of the specialized electrically isolated rooms at the Neurophysiology Department. This will be dubbed "basal recording". The equipment used is also the standard one used for routine postoperative recordings.
3. 5 days after the initial surgery, and following the protocol in place for these procedures, the tunnelization and battery placement will take place. This is done under general anaesthesia. During anaesthetic induction, the patient is exposed to incremental doses of propofol. Different plasmatic concentrations will be targeted using the mathematical model in the target controlled infusion (TCI) pump. These recordings will be called "propofol at a 0.5, 1, 1.5, 2, 2.5 μg/mL".

ELIGIBILITY:
Inclusion Criteria:

* Capacity to understand, consent and commit for the three phases of the study.
* Older than 18 years old.
* The patient is scheduled for DBS electrode placement for PD treatment by his neurologist.

Exclusion Criteria:

* Allergy or hypersensibility to dexmedetomidine or propofol
* Cardiac blockade (types 2 and 3) without an implanted pacemaker
* Low blood pressure (mean < 60 mmHg) or symptoms of low cardiac output.
* Severe cerebrovascular disease.
* Pregnancy or nursing mothers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Signal power of the local field potentials. | 5 minutes for each record
  Signal power separated in bandwidth (theta, slow beta, fast beta, gamma, high frequency); absolute and relative. The comparison will be made between the different measurements: dexmedetomidine, basal and propofol.

SECONDARY OUTCOMES:
UPDRS-III score | 2 minutes for each score
  Changes in UPDRS-III score with dexmedetomidine and propofol

CONTACTS AND LOCATIONS:
Overall Officials: Martínez S Antonio, Doctor, Principal Investigator — Staff of the deparment of Anestesiology
Locations (1):
- University of Navarra Clinic, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Krack P, Batir A, Van Blercom N, Chabardes S, Fraix V, Ardouin C, Koudsie A, Limousin PD, Benazzouz A, LeBas JF, Benabid AL, Pollak P. Five-year follow-up of bilateral stimulation of the subthalamic nucleus in advanced Parkinson's disease. N Engl J Med. 2003 Nov 13;349(20):1925-34. doi: 10.1056/NEJMoa035275. PMID 14614167
- [Background] Hamani C, Richter E, Schwalb JM, Lozano AM. Bilateral subthalamic nucleus stimulation for Parkinson's disease: a systematic review of the clinical literature. Neurosurgery. 2005 Jun;56(6):1313-21; discussion 1321-4. doi: 10.1227/01.neu.0000159714.28232.c4. PMID 15918948
- [Background] Poon CC, Irwin MG. Anaesthesia for deep brain stimulation and in patients with implanted neurostimulator devices. Br J Anaesth. 2009 Aug;103(2):152-65. doi: 10.1093/bja/aep179. Epub 2009 Jun 25. PMID 19556271
- [Background] Sassi M, Zekaj E, Grotta A, Pollini A, Pellanda A, Borroni M, Pacchetti C, Menghetti C, Porta M, Servello D. Safety in the use of dexmedetomidine (precedex) for deep brain stimulation surgery: our experience in 23 randomized patients. Neuromodulation. 2013 Sep-Oct;16(5):401-6; discussion 406. doi: 10.1111/j.1525-1403.2012.00483.x. Epub 2012 Jul 10. PMID 22780449
- [Background] Rozet I, Muangman S, Vavilala MS, Lee LA, Souter MJ, Domino KJ, Slimp JC, Goodkin R, Lam AM. Clinical experience with dexmedetomidine for implantation of deep brain stimulators in Parkinson's disease. Anesth Analg. 2006 Nov;103(5):1224-8. doi: 10.1213/01.ane.0000239331.53085.94. PMID 17056959
- [Background] Reck C, Florin E, Wojtecki L, Krause H, Groiss S, Voges J, Maarouf M, Sturm V, Schnitzler A, Timmermann L. Characterisation of tremor-associated local field potentials in the subthalamic nucleus in Parkinson's disease. Eur J Neurosci. 2009 Feb;29(3):599-612. doi: 10.1111/j.1460-9568.2008.06597.x. Epub 2009 Jan 28. PMID 19187268
- [Background] Rodriguez-Oroz MC, Lopez-Azcarate J, Garcia-Garcia D, Alegre M, Toledo J, Valencia M, Guridi J, Artieda J, Obeso JA. Involvement of the subthalamic nucleus in impulse control disorders associated with Parkinson's disease. Brain. 2011 Jan;134(Pt 1):36-49. doi: 10.1093/brain/awq301. Epub 2010 Nov 8. PMID 21059746
- [Background] Urrestarazu E, Iriarte J, Alegre M, Clavero P, Rodriguez-Oroz MC, Guridi J, Obeso JA, Artieda J. Beta activity in the subthalamic nucleus during sleep in patients with Parkinson's disease. Mov Disord. 2009 Jan 30;24(2):254-60. doi: 10.1002/mds.22351. PMID 18951542
- [Result] Rodriguez-Oroz MC, Obeso JA, Lang AE, Houeto JL, Pollak P, Rehncrona S, Kulisevsky J, Albanese A, Volkmann J, Hariz MI, Quinn NP, Speelman JD, Guridi J, Zamarbide I, Gironell A, Molet J, Pascual-Sedano B, Pidoux B, Bonnet AM, Agid Y, Xie J, Benabid AL, Lozano AM, Saint-Cyr J, Romito L, Contarino MF, Scerrati M, Fraix V, Van Blercom N. Bilateral deep brain stimulation in Parkinson's disease: a multicentre study with 4 years follow-up. Brain. 2005 Oct;128(Pt 10):2240-9. doi: 10.1093/brain/awh571. Epub 2005 Jun 23. PMID 15975946
- [Result] Venkatraghavan L, Manninen P. Anesthesia for deep brain stimulation. Curr Opin Anaesthesiol. 2011 Oct;24(5):495-9. doi: 10.1097/ACO.0b013e32834a894c. PMID 21772140
- [Result] Venkatraghavan L, Luciano M, Manninen P. Review article: anesthetic management of patients undergoing deep brain stimulator insertion. Anesth Analg. 2010 Apr 1;110(4):1138-45. doi: 10.1213/ANE.0b013e3181d2a782. Epub 2010 Feb 8. PMID 20142347
- [Result] Raz A, Eimerl D, Zaidel A, Bergman H, Israel Z. Propofol decreases neuronal population spiking activity in the subthalamic nucleus of Parkinsonian patients. Anesth Analg. 2010 Nov;111(5):1285-9. doi: 10.1213/ANE.0b013e3181f565f2. Epub 2010 Sep 14. PMID 20841416
- [Result] Steigerwald F, Hinz L, Pinsker MO, Herzog J, Stiller RU, Kopper F, Mehdorn HM, Deuschl G, Volkmann J. Effect of propofol anesthesia on pallidal neuronal discharges in generalized dystonia. Neurosci Lett. 2005 Oct 7;386(3):156-9. doi: 10.1016/j.neulet.2005.06.012. PMID 16024174
- [Result] Rozet I. Anesthesia for functional neurosurgery: the role of dexmedetomidine. Curr Opin Anaesthesiol. 2008 Oct;21(5):537-43. doi: 10.1097/ACO.0b013e32830edafd. PMID 18784476
- [Result] Elias WJ, Durieux ME, Huss D, Frysinger RC. Dexmedetomidine and arousal affect subthalamic neurons. Mov Disord. 2008 Jul 15;23(9):1317-20. doi: 10.1002/mds.22080. PMID 18442130